CLINICAL TRIAL: NCT02286752
Title: Comparison of the Effects of Neostigmine With Sugammadex on Postoperative Nausea and Vomiting.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, özgür yağan, MD, Ordu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Odu-6
Record Dates: First submitted 2014-11-03; First posted 2014-11-10 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2015-01

CONDITIONS: Incidence of Postoperative Nausea and Vomiting
MeSH Terms: conditions — Vomiting | interventions — Neostigmine; Sugammadex

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- neostigmine (Active Comparator)
  Interventions: Drug: Neostigmine
- sugammadex (Active Comparator)
  Interventions: Drug: sugammadex

INTERVENTIONS:
Drug: Neostigmine — for reversal of neuromuscular block: 0,05 mg kg-1 neostigmine + 0,025 mg kg-1 atropine
  Arms: neostigmine
Drug: sugammadex — for reversal of neuromuscular block: sugammadex 2 mg kg-1
  Arms: sugammadex

SUMMARY:
Postoperative nausea and vomiting is one of most common complications after general anesthesia. Female sex, history of postoperative nausea and vomiting, motion sickness, non smoker status, opioid administration are known as risk factors for developing postoperative nausea and vomiting.

It has been suggest that antagonism of residual neuromuscular block with a mixture of neostigmine and atropine at the end of the surgery increases the risk of postoperative nausea and vomiting.

Sugammadex is a very safe drug with almost no serious adverse effects. The known adverse effects include slight coughing, movement, an altered taste sensation in the mouth, transient prolongation of the QT interval, hypersensitivity, and a short term prolongation of the activated partial thromboplastin time.

The aim of this study was to compare the sugammadex versus neostigmine plus atropine for reversal of rocuronium induced neuromuscular blockade in terms of incidence of postoperative nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status 1 and 2
* endotracheal intubation and general anesthesia scheduled for elective surgery

Exclusion Criteria:

* age < 18 years, > 65 years
* pregnancy
* refusal to participate and patients already participating in another study
* allergy to study drugs
* communication difficulty
* psychiatric and neurological disorders
* use of analgesics or sedative or antiemetic drugs within 24 hours before surgery.
* emergency surgery
* history of drug or alcohol abuse
* ASA 3 and above
* patients with vertigo
* Laparoscopic surgery, oncologic surgery, strabismus and mid ear surgery neurosurgery, gynecologic surgery, breast surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2014-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Verbal Descriptive Scale | within postoperative 24 hours
  0: no nausea 1: mild 2: moderate 3: severe

CONTACTS AND LOCATIONS:
Locations (1):
- Anesthesiology and Reanimation Dept. Ordu University Training and Research Hospital, Altinordu, Ordu, Turkey (Türkiye)